CLINICAL TRIAL: NCT06881758
Title: High Intensity Training for Patients with Anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Martin Kragnes Bystad, Head of research, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 714458
Record Dates: First submitted 2024-12-13; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Depression Anxiety Disorder; Blood Pressure Check (Hypertension Screening)
Keywords: physical exercise; mental health; high intensity training
MeSH Terms: conditions — Anxiety Disorders; Motor Activity; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High intensity exercise training (Experimental): High intensity exercise training
  Interventions: Behavioral: Exercise
- Low intensity exercise training (Active Comparator): Low intensity exercise training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The investigators will investigate the differences between high and low intensity training

SUMMARY:
The aim of the current project is to examine the effects of high intensity exercise (by using 1x4 intervals) to reduce symptoms of anxiety in patients in mental health care. The expected benefits for patients are positive health effects, by improving physical fitness and reducing psychological symptom burden. The patients will have the opportunity to learn to use physical activity as a specific measure to be used in their own lives and be a source of coping. Furthermore, knowledge about physical activity and mental health may be applicable in mental health care as a part of a treatment plan.

DETAILED DESCRIPTION:
The study is a randomised controlled trial ("RCT") design with a 1:1 allocation into two groups. The two groups are high intensity exercise (1x4 minutes performed two times per week with a heart rate above 85% of maximal heart rate) and low intensity exercise (45 minutes performed two times per week with a heart rate of approximately 60% of maximal heart rate). The total amount of training sessions for both groups will be eight. The high intensity exercise group will serve as the intervention group, while the low intensity exercise group will serve as an active control group.

The patients will be randomly allocated (randomised) to these groups. An exercise physiologist (holding a master's degree in exercise physiology) will supervise the training sessions. The training sessions will take place in a dedicated room using a treadmill and a heart rate monitor. The training sessions will be individual.

The primary outcome measure will be degree of anxiety symptoms measured by Hospital Anxiety and Depression Scale (HADS) and Beck Naxiety Inventory (BAI) prior to the first (pre) and after the last (post) training session is completed. Secondary outcome measures will be compliance, i.e. to what degree the patient is able to sustain the exercise regimen three months after participating in the project, in addition to the patient's blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild/moderate anxiety disorders, aged 18-60 years. Anxiety disorders in accordance with F 41 in ICD-10, including generalised anxiety disorder, agoraphobia/panic disorder, social phobia, post-traumatic stress disorder, hypochondria, and obsessive-compulsive disorder.
* Comorbidity will occur, so the patient may also have depression. However, the main disorder should be anxiety.

Exclusion Criteria:

* Somatic diseases that may impede training: cardiovascular disease, severe asthma, severe COPD, cancer, poorly regulated diabetes.
* Schizophrenia or bipolar disease
* Suicidality (prior attempts or ongoing risk of suicide)
* Substance addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | HADS will be performed on the first day the patient attends the study and on the very last day the patient attends.
  Hospital Anxiety and Depression Scale (HADS). This a questionnaire generating a scale ranging from 0 to 42 points. Lower scores mean a better outcome.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | We will measure the blood pressure on the first day the patient attends the study and on the very last day the patient attends.
  Blood pressure
Beck Depression Inventory | Beck Depression Inventory will be performed on the first day the patient attends the study and on the very last day the patient attends.
  Beck Depression Inventory is a questionnaire for detecting depressive symptoms. This questionnaire range from 0 to 63. Lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to various reasons, including concerns about patient privacy and confidentiality, legal or ethical restrictions, the potential risk of re-identifying participants, and the protection of sensitive data.

REFERENCES:
- [Derived] Bystad M, Rydland S, Bugge C, Hogmo S, Brondbo B, Jacobsen R, Garcia-Fernandez L, Rodriguez-Jimenez R, Romero-Ferreiro V, Wynn R. High-intensity training vs. low-intensity training for patients with anxiety: a randomised controlled trial. Trials. 2026 Jan 27. doi: 10.1186/s13063-026-09472-2. Online ahead of print. PMID 41593737